CLINICAL TRIAL: NCT02605941
Title: DNA Methylation Biomarkers for Cervical Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: iStat Biomedical CO., Ltd. (Industry)
Collaborators: Mackay Memorial Hospital (Other); Li Shin Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: epigene-13151
Record Dates: First submitted 2015-11-06; First posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer
Keywords: DNA methylation; Cervical cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cervical cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this prospective study is to evaluate whether DNA methylation can be applied in cervical cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* women with age ≥20 and sexual experience
* Agree to sign ICF

Exclusion Criteria:

* women had received Hysterectomy
* women had destructive therapy for cervical lesions in 6 months, for examples: conization, Laser or cryotherapy, chemotherapy, and radiation therapy
* Women are at pregnancy or had baby delivery in 6 weeks

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investigators plan to recruit 5,000 women to participate this study in Taiwan. Papanicolaou test, high-risk HPV typing and DNA methylation will be co-tested. It is expected to find an optimal solution for molecular cervical cancer screening. The participant will be recruited by Mackay Memorial Hospital, Chang Gung Memorial Hospital, and Lin-Hsin Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Performance of DNA methylation in identification of CIN3 or worse. | 3 years
  Patient's information, including clinical diagnosis and the molecular testing results etc., will be collected. Performances of the screening tools will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-cheng Yang, MD, Study Chair — Mackay Memorial Hospital; Shih-chu Ho, MD, Principal Investigator — Li Shin Hospital; Ting-Chang Chang, MD., MPH., Principal Investigator — Chang Gung Memorial Hospital; Chih-Long Chang, MD, Ph.D., Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Linkou Chang Gung Memorial Hospital, Lin-Shin Medical Corporation Lin-Shin Hosptial, Taipei, Taoyuan, and Taichung, Taiwan

REFERENCES:
- [Background] Sova P, Feng Q, Geiss G, Wood T, Strauss R, Rudolf V, Lieber A, Kiviat N. Discovery of novel methylation biomarkers in cervical carcinoma by global demethylation and microarray analysis. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):114-23. doi: 10.1158/1055-9965.EPI-05-0323. PMID 16434596
- [Background] Lai HC, Lin YW, Huang TH, Yan P, Huang RL, Wang HC, Liu J, Chan MW, Chu TY, Sun CA, Chang CC, Yu MH. Identification of novel DNA methylation markers in cervical cancer. Int J Cancer. 2008 Jul 1;123(1):161-7. doi: 10.1002/ijc.23519. PMID 18398837
- [Background] Huang TH, Lai HC, Liu HW, Lin CJ, Wang KH, Ding DC, Chu TY. Quantitative analysis of methylation status of the PAX1 gene for detection of cervical cancer. Int J Gynecol Cancer. 2010 May;20(4):513-9. doi: 10.1111/IGC.0b013e3181c7fe6e. PMID 20442585
- [Background] Lai HC, Lin YW, Huang RL, Chung MT, Wang HC, Liao YP, Su PH, Liu YL, Yu MH. Quantitative DNA methylation analysis detects cervical intraepithelial neoplasms type 3 and worse. Cancer. 2010 Sep 15;116(18):4266-74. doi: 10.1002/cncr.25252. PMID 20564139
- [Background] Chao TK, Ke FY, Liao YP, Wang HC, Yu CP, Lai HC. Triage of cervical cytological diagnoses of atypical squamous cells by DNA methylation of paired boxed gene 1 (PAX1). Diagn Cytopathol. 2013 Jan;41(1):41-6. doi: 10.1002/dc.21758. Epub 2011 Jun 27. PMID 21710649
- [Background] Krane JF, Granter SR, Trask CE, Hogan CL, Lee KR. Papanicolaou smear sensitivity for the detection of adenocarcinoma of the cervix: a study of 49 cases. Cancer. 2001 Feb 25;93(1):8-15. PMID 11241260